CLINICAL TRIAL: NCT01475929
Title: Effect of Probiotic Supplement on Bowel Function
Acronym: IBS2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol violations
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IBS2
Record Dates: First submitted 2011-09-20; First posted 2011-11-22 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; probiotic
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotic low (Active Comparator): Lower dose of probiotic supplement
  Interventions: Dietary Supplement: Probiotic supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Probiotic supplement
- Probiotic high (Active Comparator): Higher dose of probiotic supplement
  Interventions: Dietary Supplement: Probiotic supplement

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — A single strain probiotic supplement given at two doses
  Other Names: Lactobacillus

SUMMARY:
The purpose of this study is to analyse the effect of probiotic supplement on symptoms of irritable bowel syndrome.

DETAILED DESCRIPTION:
The aim of the intervention is to analyse the effect of a probiotic supplement in a dose-responsive set up on symptoms of irritable bowel syndrome (IBS). Fulfillment of Rome III criteria will be used as inclusion criterion. Subjective assessment of bowel symptoms, IBS-related quality of life and adequate relief will be assessed as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 65 with functional bowel symptoms and fulfilling Rome III criteria for IBS will be recruited. Sufficient general health and orientation for participating in the study is required and will be evaluated by the MDs.

Exclusion Criteria:

* Diagnosed or suspected organic gastrointestinal diseases or severely impaired general health are exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in functional bowel symptoms | 0 weeks, 6 weeks, 12 weeks
  Validated questionnaire

SECONDARY OUTCOMES:
Change in quality of life | 0 weeks, 6 weeks, 12 weeks
  Validated questionnaire
Adequate relief | Weekly over 3 month intervention
  Weekly question
Change in faecal microbiota | 0 weeks, 6 weeks, 12 weeks
  Quantification of selected microbes and the intervention strain from faecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Ouwehand, PhD, Study Chair — Danisco; Anna Lyra, PhD, Study Director — Danisco; Lea Veijola, MD, Principal Investigator — Helsinki Health Centre; Sampo Lahtinen, PhD, Study Chair — Danisco; Anneli Tarpila, PhD, Study Director — Danisco
Locations (1):
- Herttoniemi Hospital, Helsinki, Helsinki, Finland